CLINICAL TRIAL: NCT05512234
Title: A Double-blind, Mylti-center, Randomised, Placebo-controlled, Parallel-group Study Evaluating the Effect of Probiotic Limosilactobacillus Reuteri (L. Reuteri) on Crying and Fussing Time in Infants With Colic
Brief Title: Effect of Probiotic Limosilactobacillus Reuteri (L. Reuteri) on Crying Time in Infants With Colic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0197
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Colic, Infantile
Keywords: Colic; L. reuteri
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. reuteri (Experimental): 5 drops administered once daily for 21 days
  Interventions: Dietary Supplement: L. reuteri
- Placebo (Placebo Comparator): 5 drops administered once daily for 21 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri — Dietary supplementation with drops containing L. reuteri once daily for 21 consecutive days
  Arms: L. reuteri
Dietary Supplement: Placebo — Dietary supplementation with placebo drops identical to those containing L. reuteri once daily for 21 consecutive days
  Arms: Placebo

SUMMARY:
This is a double-blind, multi-center, randomized, placebo-controlled, parallel-group study in infants with colic with the primary objective to evaluate crying time.

DETAILED DESCRIPTION:
Prevalence of infantile colic varies according to the definition used but estimates range between 5 % and 26 % of the infant population. To differentiate colic from other, more serious conditions it should be characterized by several clinical features. Infant colic is often accompanied by flushing the face, frown, tensing of the abdomen, clenching of the fists, and drawing up the leg, frequent, prolonged, and intense crying or fussiness in a healthy infant. Even though infant colic is benign and usually self-limiting condition it is a source of major distress for the infant, parents, family, and health care givers.

Despite infant colic occurs frequently, little agreement has been reached on the definition, pathogenesis, or the optimal management strategy for infant colic. Recent systematic reviews and meta-analyses showed that probiotic L. reuteri DSM 17938 supplementation significantly lowered the number of hours of crying and fussing daily. A significant peak effect was seen at 3 weeks in most studies. Interestingly, babies with infant colic were found to have increased evidence of gut inflammation, as evidenced by high levels of the antimicrobial peptide fecal calprotectin; also, the levels of fecal calprotectin declined significantly as the condition resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 3-8 weeks at screening.
2. Gestational age 37+0 weeks - 42+0 weeks at birth.
3. Birth weight appropriate for gestational age (AGA - weight between 10th and 90th percentile) or Large for Gestational Age (LGA - weight above the 90th percentile) determined using WHO Weight-for Age percentile guides.
4. Parents/caregivers/legal guardians are >18 years.
5. Exclusively or predominantly breastfed infants (> 50 % breast fed).
6. Willing to maintain current feeding patterns (not change formula/not change ratio of formula:breast milk etc.).
7. Readiness and the opportunity for parents/caregivers/legal guardians to fill out a study diary, questionnaires.
8. Infantile colic diagnosed according to Rome IV criteria (face-to-face consult with a physician, parents/caregivers/legal guardians must report that their infant has cried or fussed for 3 or more hours per day, during 3 or more days in the preceding week). At Visit 2, this will be confirmed by Baby's Day Diary®, at least one 24-hour period should show 3 or more hours of crying/fussing time.
9. Parents/caregivers/legal guardians with ability to understand and comply with the requirements of the study, as judged by the Investigator.
10. Parents/caregivers/legal guardians willing and able to give informed consent for their and their infant's participation in the study.
11. The mother of the infant must be willing to attend Visit 2 (Day 0), Visit 4 (Day 8), and Visit 6 (Day 22).
12. Infant is considered healthy, in the opinion of the investigator following physical exam.

Exclusion criteria

1. Infants with severe gastroesophageal reflux (throwing up or spitting up more than a teaspoon of milk > 8 times daily, projectile, bilious or bloody emesis).
2. Infants with failure to thrive, intrauterine growth retardation, haematochezia (blood in the stools), diarrhoea (watery stools that takes the shape of a container > 12x in breastfed and >5 in partially breastfed infants daily), or fever (38.0 degrees), as reported by parents/caregivers/legal guardians.
3. Infants with congenital heart disease, immunodeficiency, asplenia, cancer, cystic fibrosis, and those with liver disease.
4. Infants with reported exposure to probiotics in the 7 days prior to Screening Visit (V1) and throughout the study period.
5. Infants with reported exposure to oral and/or systemic antibiotics in the 7 days prior to Screening Visit (V1) and throughout the study period.
6. Infants with reported exposure to medications, therapies, or products with the aim to relieve infantile colic including proton pump inhibitors in the 7 days prior to Screening Visit (V1) and throughout the study period.

Ages: 3 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Crying and fussing time | From baseline to Day 7
  Change in daily crying and fussing time measured by Baby Day Diary

SECONDARY OUTCOMES:
Crying and fussing time | From baseline to Day 3, Day 5, Day 14, Day 21
  Change in mean daily crying and fussing time measured by Baby Day Diary
Crying time | From baseline to Day 3, Day 5, Day 7, Day 14, Day 21
  Change in mean daily crying time measured by Baby Day Diary
Number of responders | From baseline to Day 3, Day 5, Day 7, Day 14, Day 21
  Proportion of responders defined as reduction of daily average crying time with 50 % compared to baseline
Family quality of life (family QoL) | From baseline to Day 7 and Day 21
  Change in family QoL measured by the PedsQL Family Impact Module (Acute) - Total Score
Sleeping time | From baseline to Day 3, Day 5, Day 7, Day 14, Day 21
  Change in mean sleeping time measured by Baby Day Diary
Maternal depression | From baseline to Day 7 and Day 21
  Change in maternal depression measured by the Edinburgh Postnatal Depression Scale Total Score

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Palming, PhD, Study Director — BioGaia AB
Locations (2):
- Atlantia Clinical Trials, Cork, Ireland
- Clinical Trail Consultants AB, Uppsala, Sweden